CLINICAL TRIAL: NCT00828763
Title: An Open Label, Non-Randomized, Single Dose, Mass Balance Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C-GSK1349572 20 mg, Administered as a Single Oral Suspension Dose to Healthy Adult Subjects (ING111853)
Brief Title: GSK1349572 Mass Balance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Study Director, GSK
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111853
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Volunteer
Keywords: healthy volunteer; radiolabelled

ARMS (1):
- 1 (Experimental): [14C]-GSK1349572 administered as a single oral dose
  Interventions: Drug: [14c}-GSK1349572

INTERVENTIONS:
Drug: [14c}-GSK1349572 — HIV-Integrase inhibitor labelled with a carbon 14 marker

SUMMARY:
Mass balance study to determine the recovery of a single radiolabelled dose of GSK1349572 from urine and feces

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male subjects between 30 and 55 years of age.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 84 days after the dose of study medication.
* Body weight ≥ 50 kg and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete the study (minimum of 6 and a maximum of 11 nights confinement in the clinical research unit).
* A history of regular bowel movements (averaging one or more bowel movements per day).
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects who have received a total body radiation dose of greater than 5.0 mSv (upper limit of WHO category II) or exposure to significant radiation (e.g. serial x-ray or CT scans, barium meal etc) in the 12 months prior to this study.
* Any condition that could interfere with the accurate assessment and recovery of radiocarbon [14C].
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 45-100 bpm. A single repeat is allowed to determine eligibility
* ECG within protocol criteria

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
• AUC (0-t), AUC (0-∞), Cmax, tmax, λz, tlag, and t1/2 of total drug-related material (radiocarbon) in blood and plasma following oral suspension [14C]-GSK1349572 dosing. | Up to 10 days
• AUC (0-t), AUC (0-∞), Cmax, tmax, λz, tlag, CL/F, Vz/F, and t1/2 of GSK1349572 in plasma following oral suspension [14C]-GSK1349572 dosing. | Up to 10 days
• Collection of samples for use in a separate study for characterization and quantification of GSK1349572-related metabolites in plasma, urine and fecal homogenates. | Up to 10 days
Percent recovery of total radiocarbon in urine and feces | Up to 10 days

SECONDARY OUTCOMES:
• Safety and tolerability parameters, including adverse events (AEs), vital signs, ECGs, and clinical laboratory assessments. | Up to 14 days
Blood:Plasma ratio of total drug-related material (radioactivity) | Up to 10 days
Percent of total radiocarbon associated with red blood cells | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States